CLINICAL TRIAL: NCT05406531
Title: The Effectiveness of Mobile-based Psychological Interventions in Reducing Psychological Distress and Preventing Stress-related Changes in Psycho-neuroendocrine-immune Network in Breast Cancer Survivors- Randomized Controlled Trial
Brief Title: The Effectiveness of Psychological Interventions in Psycho-neuroendocrine-immune Network in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Principal Investigator, Miroslav Světlák, Department head (Department of Psychology and Psychosomatics MUNI), Masaryk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AZV2022
Record Dates: First submitted 2022-02-25; First posted 2022-06-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer Female; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Biomarkers; mHealth; psychological intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online (Experimental): MBCT-Ca uses cognitive behavioral therapy (CBT) methods in collaboration with mindfulness meditative practices and similar psychological strategies.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online
- Positive Psychology - online (Experimental): Positive psychology is focused on the character strengths and behaviors that allow individuals to build a life of meaning and purpose.
  Interventions: Behavioral: Positive Psychology - online
- Autogenic Training - online (Experimental): Autogenic training is a relaxation technique focusing on promoting feelings of calm and relaxation to help reduce stress and anxieties.
  Interventions: Behavioral: Autogenic Training - online
- Waiting list (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online
Behavioral: Positive Psychology - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Positive Psychology - online
Behavioral: Autogenic Training - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Autogenic Training - online

SUMMARY:
In this study researchers will examine an influence of three different psychological interventions in the form of mobile application on psycho-neuroendocrine-immune system among breast cancer survivors.

DETAILED DESCRIPTION:
Background:

Most studies focusing on the effects of psychological interventions on health-related outcomes have relied on self-reports. There is also growing research interest in the effects of such interventions on directly measurable biological processes associated with chronic stress. Neuroendocrine-immune system interactions are fundamental tools through which stress affects the course of cancer. The study will examine effect of three psychological interventions on most frequently studied stress related biomarkers: cortisol, HRV (heart- rate variability), CRP, relative and absolute counts of: B-lymphocytes ,T-lymphocytes, NK-cells, NK-T-like cells, monocytes; cytokine levels. Although current research suggests salutogenic changes in the immune profile of cancer patients as a result of psychological interventions, the results of individual studies are still inconsistent. To get clearer outcomes researchers decided to follow recommendations for researchers in manner that optimizes study design: to recruit very homogenous sample of cancer patients, to continue measurements in 3 and 9 months follow up, to collect data on individual´s adherence to protocol of mobile application.1,2 In addition to biomarkers, researchers will monitor changes in psychological variables.

Aims of the project and main hypotheses:

1. To test the long-term and short-term effectiveness of eHealth adaptations of three standardized mental health support programmes for cancer patients (MBCT-Ca, PP and AT) - administered through the mobile application MOÚ MindCare, in reducing psychological distress and preventing changes in the functioning of the autonomic nervous system, endocrine system and immune system that have been linked to chronic stress and are likely to have a negative impact on both mental and physical health in the long-term perspective if not managed. The investigators expect that participants in all three intervention group will show more adaptive psychological functioning, higher quality of life, lower levels of stress, depression, anxiety, fatigue, sleep disturbances and other common problems associated with breast cancer survivorship, higher HRV levels and lower cortisol levels as compared to the treatment-as-usual control group, when controlling for pre-intervention values. The investigators also expect group differences in immune system functioning, correlated with differences in other markers of stress.
2. To compare the potentially differential effects of the three intervention programmes on biological and psychological indicators of stress and quality of life. The investigators tentatively expect programmes involving a cognitive component (MBCT-Ca and PP) to be more effective than AT, especially for psychological outcomes.
3. To examine the extent to which the observed effects of each programme are mediated by characteristics the interventions are primarily expected to influence. The investigators expect the effect of MBCT to be primarily mediated by mindfulness, self-compassion and emotion regulation, and the effect of PP to be primarily mediated by self-compassion, gratitude and perceived hope.
4. To evaluate the moderating roles of intervention adherence and perceived acceptability in the effectiveness of the intervention programmes. The investigators expect higher adherence and acceptability to be associated with greater improvement in the outcome variables. These data will also help identify types of individuals for whom each programme might be most and least suitable and provide information on sources of potential problems with MOÚ MindCare - or generally mHealth - intervention adherence.

Methods:

The research is conceptualized as a randomized control trial employing a 4 × 4 factorial design. Participants will be randomly assigned to one of the four arms: 1. MBCT-Ca (Mindfulness Based Cognitive Therapy for Cancer) 2. PP (Positive Psychology) 3. AT (Autogenic training) 4.WL (Waiting list). Participants will take the 8 week online program via mobile application. Assessment measurements will be collected in four phases. Phase 1: Assessment at the start of the programme. Phase 2: Assessment in the week after programme completion. Phase 3: Follow-up assessment 3 months after the end of programme. Phase 4: Follow-up assessment 9 months after the end of programme. Data collection will contained: collection of blood samples, single lead ECG, administration of self-report measures. Main data collection points will be synchronized with regular check-ups for each participant to minimize drop-out rates and the burden on the participants.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18
* Breast cancer patients at the end of adjuvant treatment

Exclusion Criteria:

* Patients without a mobil device ("smart" mobile phone)
* Patients without internet access
* Patients with diagnosed: psychotic disorder; severe depressive episode; panic disorder; bipolar disorder; personality disorder associated with uncontrollable mood swings; PTSD; suicidal attempts and active suicidal ideation; disability pension due to non-specific mental or somatic problems; hospitalization due to a psychiatric disorder in the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) using ECG | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  HRV will be obtained from ECG measured according to a protocol involving a standardized sequence of measurements taken at rest with uncontrolled and controlled breathing. The completion of questionnaire related to rumination and impact of the cancer event before the measurement of rest ECG will serve as the priming of distress. The obtained data will be processed using the Kubios HRV Premium program- time-domain HRV parameters - RMSSD, SDNN, pNN50 and Power Spectrum density HRV parameters - LF power, HF power, and LF/HF ratio.
Change in symptoms of individual stress level using the Perceived Stress Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The questions in this scale ask about feelings and thoughts during the last month. Each question has five response options ranging in value from null to four (0=never; 1=almost never; 2=sometimes; 3=fairly often; 4=very often). To find the total raw score, sum the values of the response to each question (reverse code items 4, 5, 7a and 8). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Change in depression, anxiety and stres using the Depression, Anxiety and Stress Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Depression, Anxiety and Stress Scale (DASS-21) is a 21 items scale designed to measure depression, anxiety, and stress. The instrument comprises three subscales: the emotional states of depression, anxiety, and stress. Each question has four response options ranging in value from null to four (0= did not apply to me at all; 1= applied to me to some degree, or some of the time; 2= applied to me a considerable degree or a good part of time; 3= applied to me very much or most of the time). To find the total raw score, sum the values of the response to each question for each of subscale (scores will need to be multiplied by 2 to calculate the final score). The lowest possible raw score is 0 and the highest possible raw score is 42 for each subscale. A higher score represents more of the concept being measured.
Change in positive mental health using the Positive Mental Health Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Positive Mental Health Scale (PMHS) is a nine-item scale designed to measure positive mental health (combination of emotional, psychological, and social aspects of well-being). Each item on the questionnaire is scored from 0 (do not agree) - 3 (agree). The lowest possible raw score is 0 and the highest possible raw score is 27. A higher score represents more of the concept being measured.
Change in health-related quality of life using The Functional Assessment of Chronic Illness Therapy (FACIT)-Spiritual Well-Being (Sp) | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT)-(Sp) is composed of the FACT-General (FACT-G) and a 12-item Spiritual Well-Being scale (FACIT-Sp-12).The FACT-G (Version 4) is a 27-item compilation of general questions divided into four primary QOL subscales: Physical Well-Being (PWB; 7-items), Social/Family Well-Being (SWB; 7-items), Emotional Well-Being (EWB; 6-items), and Functional Well-Being (FWB; 7-items).Each question has five response options ranging in value from null to four (0= not at all; 1= a little bit; 2=somewhat; 3= quite a bit; 4=very much). The total FACT-G score is obtained by summing individual subscale scores (PWB + EWB + SWB + FWB). The lowest possible raw score is 0 and the highest possible raw score is 48 in Spiritual Well-Being subscales. The lowest possible raw score is 0 and the highest possible raw score is 108 in FACT-G. A higher score represents more of the concept being measured.

SECONDARY OUTCOMES:
Change in relative and absolute counts of B-lymphocytes (CD19+), T-lymphocytes, T-helper lymphocytes (CD3+ CD4+), T-cytotoxic lymphocytes (CD3+ CD8+), NK-cells (CD16+ CD56+), NK-T-like cells (CD3+ CD56+) and monocytes (CD14+) | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The counts will be obtained by flow cytometric immunophenotyping. For immunophenotyping tests will be collected peripheral blood sample (2,6 ml of K3EDTA-blood) of patients.
Change in cytokine levels | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  Cytokine levels (IL-1β, IL-2, IL-6, IL-8, IL-12, IFN-γ, TNFα, IL-17, IL-1ra, IL-4, IL-5, IL-10, TGF-β) will be analysed using the Bioplex 200 multiplex system. For cytokines levels will be collected peripheral blood sample (7,5 ml of blood without anti-coagulants for serum separation). Units of measurement: pg/ml (ng/l).
Change in serum cortisol level | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  Serum cortisol level will be determined by chemiluminescence-based immunoassay using the Cobas e 601 analyser (ROCHE Diagnostics). For serum cortisol level will be collected peripheral blood sample (7,5 ml of blood without anti-coagulants for serum separation ) between 9-11. a.m. Units of measurement: nmol / l.
Change in levels of C-reactive protein (CRP) | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  Levels of C-reactive protein (CRP) will be determined through the turbidimetric method automated on the Cobas c 501 module . For CRP level will be collected peripheral blood sample (7,5 ml of blood without anti-coagulants for serum separation).Units of measurement: mg/l.
Change in current emotional state using the Self-Assessment Manikin | every single morning during a whole 8 weeks of intervention; every single afternoon during a whole 8 weeks of intervention; every single evening during a whole 8 weeks of intervention
  Current emotional state will be assessed three times per day using three short items (Self-Assessment Manikin) directly incorporated in the MOÚ MindCare Application. The Self-Assessment Manikin (SAM) measures pleasure, arousal, and dominance. It is a non-verbal pictorial assessment technique.
Adherence to/satisfaction with the MOÚ MindCare application and intervention programme using the MOÚ MindCare Feasibility Questionnaire | week 9 from baseline
  Mobile application will be monitoring completing tasks by participants. Satisfaction with the MOÚ MindCare application will be measured by the MOÚ MindCare Feasibility Questionnaire. Questions have two, three, four or five response options ranging in value from one to two, three, four or five. A few questions have open answers options. To find the total raw score, sum the values of the response to each question (reverse code item: 4). The lowest possible raw score is 8 and the highest possible raw score is 26. A higher score represents more of the concept being measured.
Change in emotion dysregulation using the Difficulties in Emotion Regulation Scale-SF | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Difficulties in Emotion Regulation Scale Short Form (DERS-SF) is a measure used to identify emotional regulation issues. The measure covers 4 dimensions of emotional regulation: awareness and understanding of emotions; acceptance of emotions; the ability to engage in goal-directed behaviour and refrain from impulsive behaviour when experiencing negative emotions; and access to emotion regulation strategies perceived as effective. Each question has five response options ranging in value from one to five (1=almost never; 2=sometimes; 3=about half of the time; 4=most of the time; 5=almost always). The lowest possible raw score is 18 and the highest possible raw score is 90. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Five Facet Mindfulness Questionnaire-15 | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The 15-item FFMQ (FFMQ-15) measures five facets: Observing, Describing, Acting with Awareness, Non-Judging of inner experience, and Nonreactivity to inner experience. Each question has five response options ranging in value from one to five (1=never or very rarely true; 2= rarely true; 3=sometimes true; 4=often true; 5=very often or always true). To find the total raw score, sum the values of the response to each question (reverse code items 3, 4, 7, 8, 9, 13 and 14). The lowest possible raw score is 15 and the highest possible raw score is 75. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Applied Mindfulness Process Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Applied Mindfulness Process Scale (AMPS) measures the application of mindfulness practices in daily life among persons participating in mindfulness-based interventions. The measure covers three domains of applied mindfulness processes: decentering, positive emotional regulation, and negative emotional regulation. Each question has five response options ranging in value from null to four (0= never; 1= rarely; 2=sometimes; 3=often; 4=almost always). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 60. A score ranging from 0-20 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Self- Compassion Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Self-compassion Scale (SCS) is a psychometrically measurement of self-compassion. The instrument comprises six subscales: Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness and Over-identification. Each item on the questionnaire is scored from 1-5 (1=almost never, 5=almost always). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 1, 2, 4, 6, 8, 13, 16, 18, 20, 21, 24 and 25). The lowest possible raw score is 26 and the highest possible raw score is 130. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Gratitude Questionnaire Six-Item Form | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Gratitude Questionnaire-Six-Item Form (GQ-6) is a self-report questionnaire measures individual differences in the proneness to experience gratitude in daily life. Each question has seven response options ranging in value from one to seven (1= strongly disagree; 2= disagree; 3= slightly disagree; 4= neutral; 5= slightly agree; 6= agree; 7= strongly agree). To find the total raw score, sum the values of the response to each question (reverse code items 3 and 6). The- Page 4 of 7 - lowest possible raw score is 6 and the highest possible raw score is 42. A higher score represents more of the concept being measured.
Change in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Perceived Hope Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Perceived Hope Scale (PHS) is self-report questionnaire measures individual judgment about one's experience and levels of hope. Each item on the questionnaire is scored from 0-5 (0= strongly disagree, 5= strongly agree). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 30. A higher score represents more of the concept being measured.
Basic personality traits using the Big Five Inventory BFI-10 | baseline
  The Big Five Inventory-10 (BFI-10) measures the Big Five personality traits: Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. Each question has five response options ranging in value from one to five (1= disagree strongly; 2= disagree a little; 3= neither agree or disagree; 4= agree a little; 5= agree strongly). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 1,3,4,5 and 7). The lowest possible raw score is 10 and the highest possible raw score is 50. A score ranging from 2-10 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in rumination and reflection using the Rumination-Reflection Questionnaire | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Rumination Reflection Questionnaire (RRQ) measures an adaptive (self-focus) and maladaptive form (self- rumination) of self-focus or self-attention. The instrument comprises two subscales: Rumination and Reflection. Each question has five response options ranging in value from one to five (1= strongly disagree; 2= disagree; 3= neutral; 4= agree; 5= strongly agree). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 6, 9, 10, 13, 14, 17, 20 and 24). The lowest possible raw score is 24 and the highest possible raw score is 120. A score ranging from 12-60 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in impact of event using the Impact of Event Scale-Revised | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Impact of Event Scale - Revised (IES-R) measures impact of recent and specific events, and post-traumatic stress disorder symptoms. The instrument comprises three subscales: Intrusion; Avoidance and Hyperarousal. Each question has five response options ranging in value from null to four (0= not at all; 1= a little bit; 2= moderately; 3= quite a bit; 5= extremely). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 88. A scores ranging from: 0-32; 0-32 and 0-24 are obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in sleep quality using the Pittsburgh Sleep Quality Index | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality and disturbances. The instrument comprises seven subscales: subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleeping medication and daytime dysfunction. Questions have four response options ranging in value from null to three and a few questions with open answers options. To find the total raw score, sum the values of the response to each question and for each subscale separately. The sum of scores for components yields one global score. The lowest possible raw score is 0 and the highest possible raw score is 21. A higher score represents more of the concept being measured.
Change in fatigue using the Fatigue Symptom Inventory | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Fatigue Symptom Inventory (FSI) measures multiple aspects of fatigue, including its perceived severity, frequency, and interference with daily functioning. Each item on the questionnaire is scored from 0-10 (0= not at all fatigued, 10= as fatigued as I could be). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 130. A higher score represents more of the concept being measured.
The total amount of received health care using the medical documentation software (GreyFox) | month 9 post-intervention
  Number of PET, CT and MR imaging examinations, number of acute hospitalizations, the total cost of care, and the type and amount of anticancer treatment will be measured by using hospital database program called "GreyFox".
Changes in severity of somatic symptoms using the Patient Health Questionnaire 15 | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Patient Health Questionnaire (PHQ-15) measures common mental disorders and is used to assess somatic symptom severity and screen for the potential somatisation and somatoform disorders. Each question has three response options ranging in value from null to two (0= not bothered at all; 1= bothered a little; 2= bothered a lot). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 30. A higher score represents more of the concept being measured.
Change in pain medication use | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The following variables about medication will be collected: name and strength of medication; number of days in the week the medication was taken (0-7), number of taken doses per the day (0-7 and more); regularity of a medication using (options: regularly/according to need).
Change in psychiatric medication use | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The following variables about medication will be collected: name and strength of medication; condition the medication is used for (options= sleep disorder/anxiety/depression/other); number of days in the week the medication was taken (0-7); number of taken doses per the day (0-7 and more); regularity of a medication using (options: regularly/according to need).
Change in pain intensity using the Numerical Rating Scale of Pain Intensity | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  Pain intensity will be measured by the Numerical Rating Scale of Pain Intensity (NRS-I) consists of a range of numbers (0-10). The lowest number is null and represents "no pain". The highest number is ten and represents "an extreme level of pain". Respondents are asked to choose the number that best represents a level of pain intensity.
Change in dealing with pain using the Pain Self-Efficacy Questionnaire | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Pain Self-Efficacy Questionnaire is a 10-item scale designed to measure the confidence of people with ongoing pain to achieve different activities despite pain. Each item on the questionnaire is scored from 0 (not at all confident) to 6 (completely confident). The lowest possible raw score is 0 and the highest possible raw score is 60. A higher score represents more of the concept being measured.

OTHER OUTCOMES:
Socio-demographic variables | baseline
  The following socio-demographic variables will be collected: gender, age, level of education, marital status, number of children (if any), employment status, any previous experience with autogenic training, psychotherapy, meditation, or another practice of self-development (how long/ how often is one practicing such activities).

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Světlák, PhD., Study Chair — Masaryk University
Locations (1):
- Faculty of Medicine, Masaryk University, Brno, Bohunice, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanada K, Alda Diez M, Salas Valero M, Perez-Yus MC, Demarzo MM, Montero-Marin J, Garcia-Toro M, Garcia-Campayo J. Effects of mindfulness-based interventions on biomarkers in healthy and cancer populations: a systematic review. BMC Complement Altern Med. 2017 Feb 23;17(1):125. doi: 10.1186/s12906-017-1638-y. PMID 28231775
- [Background] Black DS, Slavich GM. Mindfulness meditation and the immune system: a systematic review of randomized controlled trials. Ann N Y Acad Sci. 2016 Jun;1373(1):13-24. doi: 10.1111/nyas.12998. Epub 2016 Jan 21. PMID 26799456
- [Background] Heiss S, Vaschillo B, Vaschillo EG, Timko CA, Hormes JM. Heart rate variability as a biobehavioral marker of diverse psychopathologies: A review and argument for an "ideal range". Neurosci Biobehav Rev. 2021 Feb;121:144-155. doi: 10.1016/j.neubiorev.2020.12.004. Epub 2020 Dec 9. PMID 33309905